CLINICAL TRIAL: NCT06303687
Title: Imaging Pain in a Virtual World: Neuroimaging Biomarkers for Assessing Brain Mechanisms Mediating Virtual Reality Pain Management in Children
Brief Title: VR-PAT and fNIRS to Identify CNS Biomarkers of Pain
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nationwide Children's Hospital (Other)
Responsible Party: Principal Investigator, Henry Xiang, Professor of Medicine and Center Director, Nationwide Children's Hospital
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: STUDY00003496
Record Dates: First submitted 2024-02-06; First posted 2024-03-12 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Acute Pain; Pediatric ALL; Procedural Pain; Burns
Keywords: Virtual Reality; VR; fNIRS; Pain; Biomarker; Neuroimaging
MeSH Terms: conditions — Acute Pain; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Pain, Procedural; Burns; Pain

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to either the intervention (fNIRS and VR-PAT) or the control (fNIRS and standard of care) at the first research dressing change and will then crossover to the alternative group for the second laser procedure.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- VR-PAT (Experimental): Participant wears the Pico Neo 3 Pro Eye headset and actively plays the VR-PAT game while also wearing the fNIRS, during their clinically scheduled burn dressing change.
  Interventions: Other: VR-PAT
- Control (No Intervention): Participant wears the fNIRS and can engage in standard distraction techniques, during their clinically scheduled burn dressing change.

INTERVENTIONS:
Other: VR-PAT — Virtual Reality Pain Alleviation Therapy (VR-PAT) played on a Pico Neo 3 Pro Eye device
  Other Names: Virtual Reality
  Arms: VR-PAT

SUMMARY:
This study aims to use functional near-infrared spectroscopy (fNIRS) to identify and quantify pain biomarkers during burn dressing changes and pain relief induced by virtual reality (VR).

DETAILED DESCRIPTION:
The objective of this study is to develop central nervous system (CNS) biomarkers of pain experience during inpatient pediatric (age 6-17 years) burn dressing changes and pain relief induced by virtual reality (VR). We plan to use innovative functional near-infrared spectroscopy (fNIRS) to identify and quantify the targeted CNS biomarkers. The ultimate goal of this project is to optimize the CNS biomarkers for predicting and/or monitoring response to VR-based pain reduction approaches for pain management in clinical trials.

We will collaborate through a team science model to recruit n=4 pediatric burn injury subjects to address the following three specific aims:

Aim 1: To quantify the central nervous system (CNS) responses associated with self-reported pain intensity during a standard clinical procedure (burn dressing changes).

Aim 2: To assess brain response patterns to virtual reality (VR)-based interventions for pain management.

Aim 3: To assess the degree to which objective brain measures and brain responses to VR intervention modulate objective brain markers of pain.

ELIGIBILITY:
Inclusion Criteria:

1. Being treated for acute burn injury
2. Age 6-17 years, inclusive
3. Admitted to NCH burn unit for treatment
4. Have a dressing that requires daily changes over 3 days
5. Patient and family caregivers can communicate (read and write) using English

Exclusion Criteria:

1. Any wounds that may interfere with study procedures
2. Vision, hearing, or cognitive/motor impairments preventing valid administration of study measures
3. History of motion sickness, seizure disorder, dizziness, or migraine headaches precipitated by visual auras
4. Minors in foster care, prisoners, or currently pregnant
5. Suspected child abuse
6. Unable to communicate in English

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 4 (Estimated)
Dates: Start 2026-07 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Change in brain activity | Assessed continuously throughout burn dressing changes (60 minutes) for the fNIRS study period (up to 5 days)
  Mean change of hemoglobin oxygen (HBO2) concentration between VR and Control as detected by fNIRS.

SECONDARY OUTCOMES:
Procedural pain during burn dressing changes | Assessed within 15 minutes immediately after the burn dressing change about pain experienced during the procedure
  0-10 Numerical Rating Scale (NRS) (self-reported and caregiver-reported), 0(min)-10(max), with higher score indicating worse pain. Asked for worst pain, average pain, and time spent thinking about pain. Collected in both VR and Control group.
Change in procedural anxiety | Assessed at 3 time points (30 minutes prior to procedure, immediately prior to procedure, and within 15 minutes immediately following the procedure) for each dressing change
  Modified Yale Preoperative Anxiety Scale (mYPAS) (observed by researcher), 23.33(min)-100(max), with higher scores denoting higher levels of anxiety.
Self-reported VR experience | Within 15 minutes immediately following burn dressing change when in VR-PAT group
  0-10 Numerical Rating Scale (NRS) (self-reported - VR-PAT arm only), 0(min)-10(max), with higher score meaning better outcome. Asked for degree of realism, pleasure, and satisfaction with VR.

CONTACTS AND LOCATIONS:
Overall Officials: Henry Xiang, MD, MPH, PhD, MBA, Principal Investigator — Nationwide Children's Hospital
Locations (1):
- Nationwide Children's Hospital, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No
No IPD will be shared